CLINICAL TRIAL: NCT02285816
Title: A Phase I/II Study of MG1 Maraba/MAGE-A3 (MG1MA3), With and Without Adenovirus Vaccine, With Transgenic MAGE-A3 Insertion (AdMA3) in Patients With Incurable Advanced/Metastatic MAGE-A3-Expressing Solid Tumours
Brief Title: MG1 Maraba/MAGE-A3, With and Without Adenovirus Vaccine With Transgenic MAGE-A3 Insertion in Incurable MAGE-A3-Expressing Solid Tumours
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I214
Record Dates: First submitted 2014-10-31; First posted 2014-11-07 (Estimated); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Advanced/Metastatic Solid Tumours

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (MG1MA3 virus alone) (Experimental): The starting dose of MG1MA3 will be 1 x 10^10 pfu administered by IV on day 1 and day 4.MG1MA3 dose will be escalated as per protocol.
  Interventions: Biological: MG1MA3
- Arm B- AdMA3 (vaccine prime) alone (Experimental): Six patients will receive prime AdMA3 vaccine at a dose of 1x10^10 pfu administered IM on day (-14). No dose escalation is planned.
  Interventions: Biological: AdMA3
- Arm C- AdMA3 plus MG1MA3 (prime + boost) (Experimental): Prime AdMA3 vaccine will be administered as a single dose of 1x10^10 pfu IM at day (-14) followed by dose escalation of MG1MA3 boost, IV administered on days 1 & 4 at a starting dose of 1 log below the recommended phase II dose (RP2D), as determined in Arm A of this study. MG1MA3 dose will be escalated as defined in protocol.
  Interventions: Biological: MG1MA3; Biological: AdMA3

INTERVENTIONS:
Biological: MG1MA3 — MG1MA3: Boosting component of Oncolytic Vaccine
  Other Names: MG1 Maraba/MAGE-A3
  Arms: Arm A (MG1MA3 virus alone); Arm C- AdMA3 plus MG1MA3 (prime + boost)
Biological: AdMA3 — AdMA3: Priming component of Oncolytic Vaccine
  Other Names: Adenovirus/MAGE-A3
  Arms: Arm B- AdMA3 (vaccine prime) alone; Arm C- AdMA3 plus MG1MA3 (prime + boost)

SUMMARY:
This research is being done because these viruses have been shown to shrink tumours in animals and human tumour samples by selectively killing cancer cells and creating an immune response to the tumour antigen contained in the viruses. This effect has been shown to increase when the AdMA3 virus is given first. It is not clear if this treatment will offer better results than standard treatment.

DETAILED DESCRIPTION:
The purpose of the first phase of this study (phase I) is to find the dose of a new therapy, the MG1 Maraba/MAGE-A3 (MG1MA3) virus that can be given alone and in combination with the Adenovirus/MAGE-A3 (AdMA3) virus. In the first part of the study, patients may receive the Maraba virus, the Adenovirus or both viruses. To identify the highest safe dose of the Maraba virus alone or in combination the study will start at a dose lower than the one that does not cause side effects in animals. Participants are given one or both of these therapies and are watched very closely to see what side effects they have and to make sure the side effects are not severe. If serious side effects are seen in patients at the first dose level, doses of MG1MA3 may be lowered in subsequent patients. If the side effects are not serious, then more potential participants are asked to join this study and are given higher doses. This will continue until the maximum feasible dose level is reached or one of the lower doses is found that causes serious but temporary side effects. Doses higher than that will not be given.

ELIGIBILITY:
Inclusion Criteria:

* PHASE I: Patients must have histologically confirmed, unresectable locally advanced/metastatic solid tumour with positive expression of MAGE-A3 (primary or metastatic lesion) and for which there is no known life prolonging standard therapy.
* PHASE II: Patients must have histologically confirmed, unresectable locally advanced/metastatic solid tumour with positive expression of MAGE-A3 (primary or metastatic lesion) as follows:

  1. Non-small cell lung cancer (NSCLC) specifically adenocarcinoma and squamous cell carcinoma.
  2. Breast cancer
  3. Esophageal/GEJ cancer/gastric
* In phase II patients may be treated before refractory, such as while stable post treatment response to first line therapy.
* Presence of clinically and/or radiologically documented disease. At least one site of disease must be unidimensionally measurable by CT with IV contrast as follows:

  * Chest x-ray ≥ 20 mm
  * CT scan (with slice thickness of ≤ 5 mm) ≥ 10 mm-->Longest diameter
  * Physical exam (using calipers) ≥ 10 mm
  * Lymph nodes by CT scan ≥ 15 mm -->Measured in short axis
* All radiology studies must be performed within 14 days prior to registration (within 21 days if negative).
* Patients must have at least one additional tumour mass amenable to core needle or excisional biopsy (Note FNA is not acceptable) that is not a measurable lesion that will be used as a target lesion. Patients must consent to and be willing and able to undergo at least two core needle biopsies of that lesion.
* Age ≥ 18 years
* ECOG performance status of 0 or 1
* Patients must have received at least one prior standard first line regimen for advanced or metastatic disease. The regimen may have been cytotoxic chemotherapy, targeted therapy, hormonal therapy (for e.g. anastrozole) or immunotherapy providing considered a standard first line therapy. There is no limit to the number of prior regimens but investigators and their patients should carefully consider the likelihood of benefit of an immunologic therapy in heavily pretreated patients.
* For phase II, patients may be enrolled prior to disease progression, provided they have completed their first line therapy as below and they have documented stable disease on two consecutive tumour assessments (i.e. do not have evidence of tumour regression from therapy):

  * NSCLC patients may be entered after a minimum of 4-6 cycles of first line combination chemotherapy; if the patient is >70 years a single agent regimen is acceptable. If the patient has documented EGFR or ALK mutations, treatment they may have received may include an EGFR inhibitor or ALK inhibitor as first line therapy.
  * Breast cancer patients may be entered after a minimum of 6 cycles of first line therapy.
  * Patients with metastatic/recurrent esophageal carcinoma may be entered after first line chemotherapy for metastatic disease.
* Washout period between last day of prior treatment and planned start of treatment is the longest of one of the following:

  * two weeks
  * standard cycle length of prior regimen
  * 10 half-lives for investigational drugs.
  * 30 days since last dose of ipilumumab or PR1/PDL1 therapy.
* Patients must have recovered from any treatment related toxicities prior to registration (unless grade 1, irreversible and considered not clinically significant). Progression must be documented post radiotherapy if was given to the only site of measurable disease.
* Patients may have had prior radiation therapy. A minimum of 28 days (4 weeks) must have elapsed between the last dose of radiation and date of registration (14 days for a single palliative fraction of radiation to a non-target lesion). Patients must have recovered from any acute toxic effects from radiation prior to registration (unless grade 1, irreversible and considered not clinically significant).
* Previous surgery is permitted. A minimum of 28 days (4 weeks) must have elapsed between any major surgery and date of registration (7 days for minor surgery), provided that wound healing has occurred.
* Laboratory requirements done within 7 days prior to registration:

  * WBC ≥ 3.0 x 10^9/L
  * absolute neutrophils ≥ 1.5 x 10^9/L
  * platelets ≥ 75 x 10^9/L
  * INR ≤ 1.2
  * bilirubin ≤ 1.5 x UNL (upper normal limit)
  * AST and ALT ≤ 3.0 x UNL or ≤ 5.0 x UNL if patient has liver metastases
  * serum creatinine ≤ 1.5 x UNL or creatinine clearance ≥ 60ml/min
  * serum phosphate > 0.8mMol/L (grade 0-1)
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to registration and prior to tests which are considered to be study specific
* Patients who cannot give informed consent (i.e. mentally incompetent patients, or those physically incapacitated such as comatose patients) are not to be recruited into the study. Patients competent but physically unable to sign the consent form may have the document signed by their nearest relative or legal guardian. Each patient will be provided with a full explanation of the study before consent is requested.
* Patients must be accessible for treatment and follow up. Patients registered on this trial must be treated and followed at the participating centre.
* Pre-treatment biopsy must be done within 5 working days after registration and treatment is to begin within 5 working days of the pre-treatment biopsy (max. 10 working days from registration).

Exclusion Criteria:

* Patients with a history of other active or current malignancies that require active treatment
* Patients with known symptomatic brain metastases. Patients with treated and radiologic or clinical evidence of stable brain metastases, are eligible providing that they have been stable for at least 3 months, are asymptomatic and do not require corticosteroids (must have discontinued steroids at least 1 month prior to entry).
* Patients receiving concurrent treatment with other anti-cancer therapy or other investigational agents.
* Patients who have had prior treatment with AdVAC, MG1MA3 or any MAGE-A3 targeted therapy.
* Pregnant or lactating women. Men and women of childbearing potential who do not agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of the study participation.
* Serious illness or medical condition which would not permit the patient to be managed according to the protocol, including, but not limited to:

  1. History of significant neurologic or psychiatric disorder (e.g. uncontrolled psychotic disorders) which would impair the ability to obtain consent or limit compliance with study requirements.
  2. Active uncontrolled or serious infection (viral, bacterial or fungal) or a history of opportunistic infection associated with an immunodeficient state.
  3. Significant immunodeficiency due to underlying illness (e.g. known HIV/AIDS) and/or medication (e.g. systemic corticosteroids).
  4. Known myeloproliferative disorders requiring systemic therapy.
  5. Other medical conditions that might be aggravated by study treatment.
* Patients with uncontrolled pre-existing cardiovascular conditions and/or symptomatic cardiac dysfunction.
* Patients with household contacts meeting any of the following criteria are ineligible for study entry unless alternate living arrangements can be made:

  1. Women who are pregnant or nursing an infant
  2. Children < 12 months old
  3. Anyone with significant immunodeficiency due to underlying illness (e.g. HIV/AIDS) and/or medication (e.g. systemic corticosteroids)
* Use of anti-viral medication, steroids, immunosuppressive agents (cyclosporine, interferon) or immunization (including the flu shot) within 14 days prior to registration. Use of anti-viral, anti-platelet, or anti-coagulation medication that cannot be discontinued within 14 days of enrollment.
* Patients with disease/tumour invading a major vascular structure (e.g. carotid artery), tumour related impending bowel obstruction or clinically significant and/or rapidly accumulating ascites, pericardial or pleural effusions.
* Patients with conditions likely to have resulted in splenic dysfunction (e.g. splenectomy, sickle cell anemia, radiation to the spleen ≥ 20Gy, congenital asplenism).
* Patients with ≥ grade 2 dyspnea and/or requirement for supplemental oxygen. Patients with important pulmonary disease must complete a 6 minute ambulation test with O2 states ≥ 90% to be eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-01-22 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase I: Toxicity as measured by adverse events | 3 years
  To Determine maximum feasible dose (MFD) of:
  * MG1MA3 when administered alone on day 1 & day 4 (Arm A)
  * MG1MA3 when administered on day 1 & 4 or days 1, 4, 8 &11 following immunologic priming with AdMA3 (Arm C)
  * To confirm the safety profile of AdMA3 administration (Arm B).
Phase II: Objective tumour response rate (ORR) using RECIST v1.1. | 16 weeks
  To evaluate the objective tumour response rate (ORR) using RECIST v1.1.

SECONDARY OUTCOMES:
Phase I: Number and Severity of Adverse Events in patients | 8 weeks
  To determine the safety profile of:
  * MG1MA3 when administered alone (Arm A);
  * MG1MA3 when administered on day 1 & 4 or days 1, 4, 8 &11 following immunologic priming with AdMA3 (Arm C). Adverse events will be monitored on an ongoing basis by the central office and their frequencies reported semi-annually at investigators' meetings. Toxic effects will be categorized using the CTCAE. The worst event for each patient in each category or subcategory will be described. Both events related and unrelated to treatment will be captured.
Phase I: MG1MA3 clearance and secondary replication from pharmacokinetics and viral shedding | 3 years
  To determine the pharmacokinetics, including viral shedding, of MG1MA3 when administered:
  * Alone on day 1 & day 4 (Arm A);
  * Following immunologic priming with AdMA3 (Arm C). Pharmacokinetic parameters including MG1MA3 clearance and secondary replication (genomes and infectious units), will be evaluated in blood over time and summarized descriptively by treatment arms in phase I portion.
Phase I: Delivery to, and viral detection and replication within, tumours for MG1MA3 | 3 years
  To determine the delivery to, and viral detection and replication within, tumours for MG1MA3 when administered:
  * Alone on day 1 & day 4 (Arm A);
  * Following immunologic priming with AdMA3 (Arm C).
Phase I: Cellular and humoral immune response to virus and tumour antigens | 3 years
  To determine the cellular and humoral immune response to virus and tumour antigens (for all arms).
Phase I: Efficacy using RECIST v1.1 and iRECIST | 3 years
  To evaluate preliminary evidence of efficacy using RECIST v1.1 and iRECIST
Phase II: pharmacokinetics (PK) of MG1MA3 (MG1MA3 clearance and secondary replication (genomes and infectious units) | 3 years
  To further explore the pharmacokinetics (PK) of MG1MA3. Pharmacokinetic parameters including MG1MA3 clearance and secondary replication (genomes and infectious units), will be evaluated in blood over time and summarized descriptively by tumour types in phase II portion.
Phase II: cellular and humoral immune response to virus and tumour antigens | 16 weeks
  To further evaluate the cellular and humoral immune response to virus and tumour antigens.
Phase II: toxicity as measured by adverse events of MG1MA3 following AdMA3 | 3 years
  To further explore the safety profile of MG1MA3 following AdMA3
Phase II: Response by iRECIST | 16 weeks
  To evaluate response by iRECIST

CONTACTS AND LOCATIONS:
Overall Officials: Derek Jonker, Study Chair — Ottawa Hospital Research Institute
Locations (4):
- Canada (4):
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mullins-Dansereau V, Myre ML, Bardoul A, Geoffroy K, Rallo Pita MJ, Beland D, Desaulniers KL, Roy DG, Bourgeois-Daigneault MC. Oncolytic VSV-IL-2 has enhanced anticancer vaccination adjuvant abilities. J Immunother Cancer. 2025 May 19;13(5):e010570. doi: 10.1136/jitc-2024-010570. PMID 40389376
- [Derived] Jenner AL, Cassidy T, Belaid K, Bourgeois-Daigneault MC, Craig M. In silico trials predict that combination strategies for enhancing vesicular stomatitis oncolytic virus are determined by tumor aggressivity. J Immunother Cancer. 2021 Feb;9(2):e001387. doi: 10.1136/jitc-2020-001387. PMID 33608375
- [Derived] Pol JG, Acuna SA, Yadollahi B, Tang N, Stephenson KB, Atherton MJ, Hanwell D, El-Warrak A, Goldstein A, Moloo B, Turner PV, Lopez R, LaFrance S, Evelegh C, Denisova G, Parsons R, Millar J, Stoll G, Martin CG, Pomoransky J, Breitbach CJ, Bramson JL, Bell JC, Wan Y, Stojdl DF, Lichty BD, McCart JA. Preclinical evaluation of a MAGE-A3 vaccination utilizing the oncolytic Maraba virus currently in first-in-human trials. Oncoimmunology. 2018 Sep 19;8(1):e1512329. doi: 10.1080/2162402X.2018.1512329. eCollection 2019. PMID 30546947